CLINICAL TRIAL: NCT00476658
Title: Characterisation of Macrophage Infiltration in Obesity and Its Complications
Brief Title: Macrophage Infiltration in Human Adipose Tissue
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P050318
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2007-05

CONDITIONS: Obesity; Diabetes
Keywords: Obesity; macrophage infiltration; insulinoresistance; inflammation
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — adipose tissue, visceral adipose tissue, muscle, liver, bowel and stomach
Oversight: Data Monitoring Committee: No

SUMMARY:
Quantification of macrophage infiltration and characterization of macrophage phenotype in adipose tissue of 60 obese subjects and 20 non obese subjects

DETAILED DESCRIPTION:
Obesity results from a disequilibrium in energy balance and an inability to adapt to lifestyles which encourage increased energy intake and sedentariness. These last years, numerous studies contributed to show that obesity is the pathology of an organ, the white adipose tissue (AT), characterized by a low grade inflammation when it is enlarged. The fact that adipocytes secrete a number of inflammatory factors or "adipokines" has forced several groups to reassess the involvement of the AT in wide range of physiological and pathophysiological processes. Adipose tissue probably contributes to the links between obesity, inflammation and insulin-resistance. Our previous results based on transcriptomics studies, showed that genes encoding inflammatory molecules are mobilized in adipose tissue of obese subjects and that caloric restriction improves greatly inflammatory profile. Our preliminary studies on the morphology of adipose tissue lead us to observe a major infiltration of macrophages in morbidly obese subjects. This project is based on a clinical protocol performed in massively obese subjects (BMI>40 kg/m²), where drastic weight loss is achieved by gastric bypass. This project has several objectives. It will allow us to characterize the infiltration of macrophages in the subcutaneous adipose tissue of 60 obese subjects compared with 20 normal-weight subjects, to study the evolution during surgically-induced weight loss and to compare the infiltration observed in adipose tissue to that of other tissues (visceral adipose tissue, muscle, liver, bowel and stomach). This study will be not only quantitative (number of macrophages) but also qualitative by characterizing the phenotype of macrophages with transcriptomics and immunohistochemical approaches. We will analyze the relationships between morphological characteristics of adipose tissue and clinical and biochemical parameters related to insulin sensitivity. More generally, this project might lead us to go thoroughly into the knowledge of the link between obesity and associated comorbidities, particularly metabolic complications, and to consider novels therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Obese subjects group :

  * Obesity with BMI> 40 kg/m² or obesity with BMI between 35 and 40 kg/M² with comorbidities (OAS, diabetes, hypertension etc…)
  * Age: 18-60
* Non obese subjects group

  * Abdominal surgery planned
  * Age: 18-60

Exclusion Criteria:

* Inflammatory disease
* cancer
* stroke
* Drugs (AINS)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Inclusion Criteria:
  * Obese subjects group :
    * Obesity with BMI> 40 kg/m² or obesity with BMI between 35 and 40 kg/M² with comorbidities (OAS, diabetes, hypertension etc…)
    * Age: 18-60
  * Non obese subjects group
    * Abdominal surgery planned
    * Age: 18-60
  Exclusion Criteria:
  * Inflammatory disease
  * cancer
  * stroke
  * Drugs (AINS)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine POITOU-BERNERT, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- APHP Hopital Hotel Dieu, Paris, France

REFERENCES:
- [Derived] Bel Lassen P, Nori N, Bedossa P, Genser L, Aron-Wisnewsky J, Poitou C, Surabattula R, Juul Nielsen M, Asser Karsdal M, Julie Leeming D, Schuppan D, Clement K. Fibrogenesis Marker PRO-C3 Is Higher in Advanced Liver Fibrosis and Improves in Patients Undergoing Bariatric Surgery. J Clin Endocrinol Metab. 2022 Mar 24;107(4):e1356-e1366. doi: 10.1210/clinem/dgab897. PMID 34905051
- [Derived] Sell H, Poitou C, Habich C, Bouillot JL, Eckel J, Clement K. Heat Shock Protein 60 in Obesity: Effect of Bariatric Surgery and its Relation to Inflammation and Cardiovascular Risk. Obesity (Silver Spring). 2017 Dec;25(12):2108-2114. doi: 10.1002/oby.22014. Epub 2017 Oct 11. PMID 29024428
- [Derived] Reggio S, Rouault C, Poitou C, Bichet JC, Prifti E, Bouillot JL, Rizkalla S, Lacasa D, Tordjman J, Clement K. Increased Basement Membrane Components in Adipose Tissue During Obesity: Links With TGFbeta and Metabolic Phenotypes. J Clin Endocrinol Metab. 2016 Jun;101(6):2578-87. doi: 10.1210/jc.2015-4304. Epub 2016 Apr 6. PMID 27049236
- [Derived] Poitou C, Dalmas E, Renovato M, Benhamo V, Hajduch F, Abdennour M, Kahn JF, Veyrie N, Rizkalla S, Fridman WH, Sautes-Fridman C, Clement K, Cremer I. CD14dimCD16+ and CD14+CD16+ monocytes in obesity and during weight loss: relationships with fat mass and subclinical atherosclerosis. Arterioscler Thromb Vasc Biol. 2011 Oct;31(10):2322-30. doi: 10.1161/ATVBAHA.111.230979. Epub 2011 Jul 28. PMID 21799175
- [Derived] Dalmas E, Rouault C, Abdennour M, Rovere C, Rizkalla S, Bar-Hen A, Nahon JL, Bouillot JL, Guerre-Millo M, Clement K, Poitou C. Variations in circulating inflammatory factors are related to changes in calorie and carbohydrate intakes early in the course of surgery-induced weight reduction. Am J Clin Nutr. 2011 Aug;94(2):450-8. doi: 10.3945/ajcn.111.013771. Epub 2011 Jun 15. PMID 21677057